CLINICAL TRIAL: NCT05461599
Title: Feasibility and Acceptability of a Digital Therapeutic for Adolescent Depressive Symptoms in Cardiology and Gastroenterology
Brief Title: Digital Therapeutic for Adolescent Depressive Symptoms in Cardiology and Gastroenterology
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment too low
Sponsor: Limbix Health, Inc. (Industry)
Collaborators: Children's Hospital Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LMX-003
Record Dates: First submitted 2022-04-29; First posted 2022-07-18 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Depressive Symptoms; Major Depressive Disorder; Depression; Cardiology; Gastrointestinal Diseases; Depressive Disorder; Depressive Episode; Adolescent Behavior; Adolescent - Emotional Problem
Keywords: Depression; Mental Health; Adolescent Depression
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Gastrointestinal Diseases; Depressive Disorder; Adolescent Behavior; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- SparkRx Mobile App (Other): The 5-week SparkRx app is divided into 5 levels intended to be completed weekly. A character called 'Limbot' is used as a guide. Limbot encourages the user in completing the behavioral activation program and provides personal examples of how they have undertaken behavioral activation therapy. Participants are instructed to complete a weekly Patient Health Questionnaire (PHQ)-8 assessment and Participant Symptom Check (PSC) questionnaire in the mobile app. Tasks in the mobile app progress in a linear fashion-- i.e., each task must be completed to progress to the next task. Certain on-demand resources can be accessed in the app at any time, including crisis resources. Text entries that match a database of concerning words/phrases will trigger an automated pop-up suggesting participants visit the in-app crisis resources if they need additional support.
  Interventions: Device: SparkRx Mobile App

INTERVENTIONS:
Device: SparkRx Mobile App — The SparkRx app will be fully self-guided and completed by participants at home. It is designed to be completed over 5 weeks but users may progress through the app at their own pace. The app progresses linearly, i.e., a task must be completed before a participant can progress to the next task. Content for a given week is not expected to take more than 60 minutes to complete.

SUMMARY:
The primary aim of this pilot study is to assess the feasibility, acceptability, and preliminary evidence of efficacy of a self-guided, cognitive behavioral therapy (CBT)-based mobile app intervention (SparkRx) for symptoms of depression among adolescents being treated in specialty medical care settings at Children's Hospital of Los Angeles (CHLA).

DETAILED DESCRIPTION:
Self-report assessments will be collected at pre, post and 1-month follow up time points. Weekly PHQ-8 assessments will also be collected during the 5-week intervention as well as at pre, post and 1- month follow up time points.

Study aims involve evaluating:

* Feasibility of recruiting and enrolling adolescents with elevated symptoms of depression from the Cardiology and Gastroenterology programs at CHLA.
* Retention, program adherence, completion, and withdrawal rates.
* Safety of the intervention, including reported adverse and serious adverse events
* Perceived utility, usability, and enjoyment of the SparkRx app by adolescents
* Clinically significant changes in pre- to -post treatment depressive symptoms and persistence of such gains at 1 month follow up.

ELIGIBILITY:
Inclusion Criteria:

* 13-22 years of age at time of enrollment
* Moderate-severe self-reported symptoms of depression at baseline (PHQ-8 >=5)
* Under the care of a US-based healthcare provider and willing and able to provide the name and contact information of the provider during consent
* English fluency or proficiency and literacy of adolescent and consenting legal guardian, if required
* Access to an eligible mobile device (capable of installing the app) and regular internet access
* Willing to provide informed e-consent/assent and have legal guardian willing to provide informed e consent (if required)

Exclusion Criteria:

* Change in concurrent treatment (medication, and/or psychotherapy) for depression 30 days prior to study enrollment
* Suicide attempt within the past year
* Active suicide ideation with intent
* Previously participated in user testing or clinical testing of the Spark app
* Any condition, comorbidity, or event that, in the opinion of the investigator, will prevent the participant from adhering to the protocol or benefitting from the treatment (e.g., unable to perform informed assent or consent, treatment resistance as determined by investigator) or will prevent investigators from being able to ensure safety (e.g., will be leaving the country during study time period)

Ages: 13 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
Feasibility of intervention - Eligibility | Screening
  Percent of potential participants eligible to participate
Feasibility of intervention - Participant willingness | Screening
  Percent of eligible participants willing to participate
Feasibility of intervention - Adherence | 5 weeks
  Adherence to program: percent of enrolled participants completing all modules by post-treatment
Participant satisfaction with the SparkRx app | 5 weeks
  Acceptability of intervention. Measured by the User Experience (UXR) questionnaire. Includes questions from the UMUX-Lite; a two-item questionnaire that assesses the usability of the mobile application. Questions have seven response options from Strongly agree to Strongly disagree. Includes questions from the HaTs questionnaire; an open-ended questionnaire that assesses respondents' experiences with the product and provides options for feedback.

SECONDARY OUTCOMES:
Change in depressive symptoms | Change from screening to post-intervention (5 weeks)
  Measured by the Patient Health Questionnaire (PHQ-8). Score range of 0 to 24 with higher scores indicating worse outcome.
  * Clinically significant improvement: reduction in assessment score >= 5
  * Treatment response: 50% reduction in symptoms from pre to post-intervention
  * Remission is defined as a score < 5
Change in participant-reported health-related quality of life | Change from screening to post-intervention (5 weeks)
  Measured by the Pediatric Quality of Life Enjoyment and Satisfaction Questionnaire (PQ-LES-Q).A 15-item self-administered questionnaire that captures life satisfaction over the past week. Score range of 14 to 84 with a higher score indicating better outcome.
Change in legal-guardian reported health-related quality of life | Change from screening to post-intervention (5 weeks)
  Measured by the Pediatric Quality of Life Enjoyment and Satisfaction Questionnaire (PQ-LES-Q).A 15-item self-administered questionnaire that captures life satisfaction over the past week. Score range of 14 to 84 with a higher score indicating better outcome.
Change in participant-rated anxiety symptoms | Change from screening to post-intervention (5 weeks)
  Measured by the Generalized Anxiety Disorder scale (GAD-7).The GAD-7 is a brief 7-item assessment for generalized anxiety disorder with satisfactory sensitivity and specificity. Score range of 0 to 21 with a higher score indicating worse outcome.
Change in legal guardian-reported depressive symptoms | Change from screening to post-intervention (5 weeks)
  Measured by the Patient Health Questionnaire (PHQ-8). Score range of 0 to 24 with higher scores indicating worse outcome.
  * Clinically significant improvement: reduction in assessment score >= 5
  * Treatment response: 50% reduction in symptoms from pre to post-intervention
  * Remission is defined as a score < 5
Average treatment related usability rating | 5 weeks
  Measured by the System Usability Scale (SUS). The SUS consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree. Score range of 0 to 100 with a higher score indicating a better outcome.
Average treatment related engagement rating | 5 weeks
  Measured by the User Engagement Scale (UES-SF).A statistically reliable measure of self-reported user engagement. The form has 12 items and uses a 5 point Likert scale. Score range of 1-5 with a higher score indicating a better outcome.
Average treatment related program adherence | 5 weeks
  Measured by mobile app analytics
Average treatment related program engagement | 5 weeks
  Measured by mobile app analytics

OTHER OUTCOMES:
Health care utilization | 5 weeks
  Measured by the Healthcare Utilization Questionnaire. A two-item questionnaire that asks whether participants' have used healthcare resources in the past week.
Treatment related changes by physical symptom severity | 5 weeks
  Measured by the Functional Disability Inventory a fifteen-item questionnaire that measures functional disability and evaluates the impact of illness on the respondents' physical and psychosocial functioning in everyday social roles. Each question is rated on a 5-point scale from 0(No Trouble) to 4 (Impossible). Score range is 0 to 60 with higher scores indicating a worse outcome.
Treatment related perceptions of participants' experiences in general with SparkRx | 5 weeks
  Measured by the User Experience (UXR) questionnaire. Includes questions from the Usability Metric for User Experience-Lite; a two-item questionnaire that assesses the usability of the mobile application. Questions have seven response options from Strongly agree to Strongly disagree. Includes questions from the Happiness Tracking Surveys; an open-ended questionnaire that assesses respondents' experiences with the product and provides options for feedback.
Caregiver burden | 5 weeks
  Measured by the work absenteeism questionnaire, containing qualitative and quantitative questions about caregiving responsibilities and related impacts on employment. Higher scores are equal to more time missed from work.

CONTACTS AND LOCATIONS:
Overall Officials: Aarthi Padmanabhan, PhD, Principal Investigator — Limbix Health
Locations (1):
- Limbix Health Inc., San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No